CLINICAL TRIAL: NCT00158106
Title: Assessing the Effectiveness of Communication Therapy in the North West (The ACT NoW Pilot Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Health Technology Assessment Programme (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: HTA ref. 02/11/04; ISRCTN78617680; 04/MRE03/30
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-09

CONDITIONS: Speech or Language Impairment Following Stroke
Keywords: functional communicative ability; cost effectiveness; service user preferences
MeSH Terms: conditions — Speech | interventions — Language Therapy

INTERVENTIONS:
Procedure: Speech and Language therapy for dysarthria and/or aphasia

SUMMARY:
This study investigates the effectiveness and cost-effectiveness of speech and language therapy for adults who suffer communication difficulties following a stroke.

DETAILED DESCRIPTION:
Research Question: This is the pilot phase of a two-phase study. Phase 1 - What is the feasibility of conducting a randomised controlled trial of therapy for adults with post-stroke communication impairment? to be followed in 2006 by Phase 2 - What are the effectiveness, costs and service user preferences, for the provision of speech and language therapy for communication difficulties experienced by people in hospital with a stroke? Methodology: Phase 1 - Qualitative (focus groups & individual interviews) and quantitative (pilot RCT). Phase 2 - Qualitative (focus groups & individual interviews) and quantitative (a pragmatic, multicentred, randomised controlled trial, stratified by diagnosis and therapist/centre, using an 'intention to treat' approach). Discrete choice experiments will be used to determine cost effectiveness.

Outcome Measures: The primary outcome will be functional communicative ability. The economic analysis will estimate the incremental cost effectiveness and net benefit of the intervention group compared to the control group from a societal perspective. The qualitative study will examine service users' and carers' perspectives on the process and effects of Speech and Language Therapy or the control treatment.

Sample Group: Adults with dysarthria or aphasia, seen early after admission to hospital with a stroke. Exclusions: subarachnoid haemorrhage, progressive dementia, expected recovery without therapy.

ELIGIBILITY:
Inclusion Criteria:

* Adults with communication impairment following a new stroke

Exclusion Criteria:

* Not fluent in the English language
* Subarachnoid haemorrhage
* Pre-existing, progressive dementia or learning disability
* Palliative care only or deceased since admission
* Resident outside the treatment area

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-02; Study Completion 2005-08

PRIMARY OUTCOMES:
The primary outcome will be functional communicative ability.

SECONDARY OUTCOMES:
The economic analysis to estimate incremental cost effectiveness and net benefit of the intervention. Qualitative study to examine service users' and carers' perspectives Speech and Language Therapy vs control treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey Bowen, PhD, Principal Investigator — The University of Manchester, UK
Locations (1):
- Human Communication and Deafness, School of Psychological Sciences, Humanities Devas Street, The University of Manchester, Manchester, United Kingdom